CLINICAL TRIAL: NCT04573816
Title: Development of a Tele-monitoring Program for Patients Undergoing Surgery for Pheochromocytoma and / or Paraganglioma
Acronym: e-PPGL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: D20170803; 2020-A00144-35 (Other: IDRCB)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: follow-up; recurrence; e-consultation; Pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Use of an internet plateform — Use of an internet platform for remote monitoring of patients.

SUMMARY:
Pheochromocytomas and paragangliomas (PPGL) are rare tumors treated by surgical excision. During follow-up, more than 15% of patients will have recurrences in the form of new tumors, locoregional recurrence or metastases. This subgroup is initially not identifiable. It is therefore usual to perform annual monitoring of all patients throughout their lives by questioning and measuring blood pressure during a medical consultation and by measuring urinary or plasma metanephrines and normetanephrines.

The main objective of this prospective monocentric study is to evaluate the reliability of an optimized remote monitoring program in comparison to a usual in-clinic monitoring of patients surgically-cured and tumor-free at the time of inclusion.

DETAILED DESCRIPTION:
Patients will be included in a follow-up consultation or during a telephone contact prior to a consultation.

The period of follow-up by internet and the date of the next consultation will be fixed. This assessment is annual according to current recommendations. In the two months prior to the consultation, patients will fill out a questionnaire and transcribe their blood pressure self-measurement results as well as their biological assessment on a dedicated, approved data-hosting platform (internet application named HERMES). During the consultation, these items will be collected again without the knowledge of the results entered by the patient on the data hosting site.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Follow-up after surgery of a pheochromocytoma or a paraganglioma at the European Hospital Georges Pompidou (Paris, France)
* Free from recurrences and / or metastases at inclusion
* Non-opposition of participation in research

Exclusion Criteria:

* Lack of internet access
* Patient not understanding French
* Patient living abroad, unable to come for consultation
* Patient with co-morbidity involving life threatening within one year of inclusion
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pheochromocytoma or paraganglioma surgery
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Reliability of the program | 13 months
  Proportion of patients with a concordance score greater than or equal to 85% between the data collected in consultation and those entered by the patient via the optimized remote monitoring program

SECONDARY OUTCOMES:
Reminders | 13 months
  Evaluate feasibility of the ability of patients to actively participate in their care pathway (self care; self monitoring): number of reminders.
Schedule compliance | 13 months
  Evaluate feasibility of the ability of patients to actively participate in their care pathway (self care; self monitoring): compliance with planned deadlines.
Data filling | 13 months
  Evaluate feasibility of the ability of patients to actively participate in their care pathway (self care; self monitoring): completion of questionnaires (clinical data, blood pressure measurement and biological results).
Acceptability | 13 months
  Evaluate patient acceptability and satisfaction with the use of the solution using a satisfaction questionnaire.
Lost to follow-up | 37 months
  Establishment of an e-cohort study to evaluate the rate of patients lost to follow-up compared to the historical cohort.
Prognostic factors for recurrence. | 37 months
  Establishment of an e-cohort study to look for prognostic factors for recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence AMAR, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team.Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation(GDPR).

REFERENCES:
- [Background] Amar L, Fassnacht M, Gimenez-Roqueplo AP, Januszewicz A, Prejbisz A, Timmers H, Plouin PF. Long-term postoperative follow-up in patients with apparently benign pheochromocytoma and paraganglioma. Horm Metab Res. 2012 May;44(5):385-9. doi: 10.1055/s-0031-1301339. Epub 2012 Feb 20. PMID 22351478
- [Background] Plouin PF, Amar L, Dekkers OM, Fassnacht M, Gimenez-Roqueplo AP, Lenders JW, Lussey-Lepoutre C, Steichen O; Guideline Working Group. European Society of Endocrinology Clinical Practice Guideline for long-term follow-up of patients operated on for a phaeochromocytoma or a paraganglioma. Eur J Endocrinol. 2016 May;174(5):G1-G10. doi: 10.1530/EJE-16-0033. PMID 27048283